CLINICAL TRIAL: NCT02529605
Title: Relative Bioavailability of Two Different Milk Thistle Formulations: A Single Dose Randomized Crossover Pharmacokinetic Study
Brief Title: Relative Bioavailability of Two Different Milk Thistle Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Isagenix International LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201500360
Record Dates: First submitted 2015-08-17; First posted 2015-08-20 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Healthy
Keywords: dietary supplement; pharmacokinetics; Healthy Volunteers
MeSH Terms: interventions — milk-thistle extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Product B® IsaGenesis®, Then IsaGenesis® (Active Comparator): Participants will come into the clinic in a fasting state to receive the Product B® IsaGenesis®, which will be a one time dose of the liquid-gel formulation contained in 2 capsules, 1280 mg per capsule. After a washout period of 7 days, they will then come back to the clinic in a fasting state to receive the IsaGenesis®. This will be given for a comparison in a one time dose of the dried powder extract contained in 2 capsules; 1070 mg per capsule.
  Interventions: Dietary Supplement: Product B® IsaGenesis®; Dietary Supplement: IsaGenesis®
- IsaGenesis®, Then Product B® IsaGenesis® (Active Comparator): Participants will come into the clinic in a fasting state to receive the IsaGenesis®, which will be a one time dose of the dried powder extract contained in 2 capsules; 1070 mg per capsule. After a washout period of 7 days, they will then come back to the clinic in a fasting state to receive the Product B® IsaGenesis®. This will be given for a comparison in a one time dose of the liquid-gel formulation contained in 2 capsules; 1280 mg/capsule.
  Interventions: Dietary Supplement: Product B® IsaGenesis®; Dietary Supplement: IsaGenesis®

INTERVENTIONS:
Dietary Supplement: Product B® IsaGenesis® — This will be a crossover comparison of a one time dose of the liquid-gel formulation contained in 2 capsules; 1280 mg/capsule.
  Other Names: milk thistle extract
Dietary Supplement: IsaGenesis® — This will be a crossover comparison of a one time dose of the dried powder extract contained in 2 capsules; 1070 mg /capsule.
  Other Names: milk thistle extract

SUMMARY:
This is a single dose, randomized, cross-over pharmacokinetic study in healthy volunteers (n=12) of two dietary supplement formulations. The Product B® IsaGenesis® formulation represents a newer reformulation of an existing product known simply as IsaGenesis®. Beyond some changes in the relative abundance of some of the constituents of the earlier IsaGenesis® formulation, the Product B® IsaGenesis® product has been formulated as a liquid-gel formulation (rather than a dried powder extract) which is theorized to enhance the absorption and bioavailability of the contained botanical constituents. The purpose of this study is to compare the two dietary supplement formulations relative to the absorption of two compounds contained within the supplement known as the flavonolignans silybin A and silybin B into the bloodstream after oral administration of capsules.

DETAILED DESCRIPTION:
The study involves a total of five (5) visits to the University of Florida Shands CRC located in the Clinical Translational Research Building in Gainesville, and is expected to last approximately 6 weeks.

Screening / Informed Consent:

The Screening Visit will be conducted in the CRC and is expected to last approximately 1 hour.

After obtaining written Informed Consent, study subjects will be interviewed about their medical history and the protocol's Inclusion/Exclusion criteria will be discussed. All potential participants must be nonsmokers, not taking prescription or over-the-counter medications or botanical/nutritional supplements (inclusive of vitamins). Additionally, participants are requested to abstain from alcohol use 24 hours prior to the study health screen lab work or any scheduled study visit should they participate fully in the study.

During this initial visit, interested subjects will have blood samples drawn for health screening purposes including baseline serum chemistries, complete blood count, urinalysis, and a urine pregnancy test (women) which will precede a subsequently scheduled physical exam and possible study participation. Copies of the laboratory results will be made available to study subjects at their request. Lastly, a 12-lead electrocardiogram will be obtained.

Study Visits The following section describes the study procedures for the two major study visits at the CRC following Informed Consent and a satisfactory medical screening.

Following an overnight fast (abstention from eating any food items after 9 pm in the evening prior to the scheduled visit), subjects will arrive at the CRC the morning of the active Study Days where they will remain for approximately 8 hours on each day. After checking in, and under medical supervision, skilled CRC staff will place an indwelling venous catheter in each subject's arm to facilitate serial blood sampling. Female subjects will provide a urine sample for a pregnancy test. At approximately 8:00 AM subjects will be administered 2 capsules of either Product B® IsaGenesis® (2 capsules; 1280 mg per capsule) or IsaGenesis® (2 capsules; 1070 mg per capsule) depending on the randomization sequence assigned by the Investigational Pharmacy Services. Capsules will be administered with 240 ml of room temperature water which the subjects will be asked to drink in its entirety. Subjects will remain in a fasted state for 4 additional hours following administration of either formulation to eliminate any potential effect of food on absorption. Standard meals will be served to all subjects at least 4 hours post-dosing. The composition and amount of food eaten throughout the day will be recorded.

Blood sample collection and processing will be done by an indwelling venous catheter to facilitate serial blood sampling, a total of 9 blood samples (~10 ml each) will be taken over an 8-hour period during each of the two primary study days. Specific time points of blood collection will be immediately prior to the dose (0 time point), of either Product B® IsaGenesis® (2 capsules; 1280 mg per capsule) or IsaGenesis® (2 capsules; 1070 mg per capsule) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours.

This single dose assessment of the Product B® IsaGenesis® (2 capsules; 1280 mg per capsule) or IsaGenesis® (2 capsules; 1070 mg per capsule) pharmacokinetics will be conducted with each of the two described formulations as a single dose assessment in a randomized crossover fashion. Following the completion of the initially product administration and sample collection, a minimum 7-day wash-out period will occur prior to scheduling each subject's return for the assessment of the alternate product (under identical study conditions and collection times).

Study Exit Visit The investigators will have the subjects return within 7 days of completing the second study formulation pharmacokinetics assessment to have "exit" follow-up lab work consisting of a basic serum chemistry panel and CBC as well as urinalysis.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Race or ethnicity: no restrictions
* Body Mass Index (BMI) between 18.5 to 28 kg/m2 (inclusive)
* Satisfactory completion of the screening medical history, physical exam, and laboratory evaluations.
* Females of child-bearing potential must have a negative urine pregnancy test prior to enrollment and avoid pregnancy during study participation.
* With the exception of oral contraceptives, subjects must not be taking prescription or over the counter medication for the duration of study participation
* Subjects must have no ongoing use of any botanical/nutritional supplement, vitamin, or energy drink for the duration of study participation

Exclusion Criteria:

* The presence of a known allergy to ragweed and related plants from the Asteraceae/Compositae plant family. Members of this family include ragweed, chrysanthemums, marigolds, daisies, and some others. Milk thistle may cause an allergic reaction in people who are sensitive to these plants.
* A history (within the past year) or presence of clinically significant cardiovascular, cerebrovascular, renal, hepatic, gastrointestinal, pulmonary, immunological, hematological, endocrine, or neurologic disease will render subjects ineligible for the study.
* The presence of any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion including;

  * Gastric bezoar
  * Swallowing disorders
  * Strictures
  * Fistulas
  * GI obstruction
  * Severe dysphagia
  * Crohn's disease
  * Diverticulitis
* A positive urine pregnancy test.
* Any concomitant prescription medication, over-the-counter medication, herbal or other supplements, and vitamins during the study period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of Product B® IsaGenesis® versus IsaGenesis® | 0.0, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose
Peak Plasma Concentration (Cmax) of Product B® Isagenesis® versus IsaGenesis® | 0.0, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose

SECONDARY OUTCOMES:
Number of Participants With Response to Product B® Isagenesis® versus IsaGenesis® | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John S Markowitz, Pharm.D., Principal Investigator — University of Florida
Locations (1):
- Uf Ctsi Crc, Gainesville, Florida, United States

REFERENCES:
- [Derived] Li WY, Yu G, Hogan RM, Mohandas R, Frye RF, Gumpricht E, Markowitz JS. Relative Bioavailability of Silybin A and Silybin B From 2 Multiconstituent Dietary Supplement Formulations Containing Milk Thistle Extract: A Single-dose Study. Clin Ther. 2018 Jan;40(1):103-113.e1. doi: 10.1016/j.clinthera.2017.11.013. Epub 2017 Dec 19. PMID 29273470